CLINICAL TRIAL: NCT04054011
Title: Safety and Efficacy of Deoxycholic Acid Injection for Reduction of Upper Inner Thigh Fat
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Arisa Ortiz, Assistant Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 181524
Record Dates: First submitted 2019-06-21; First posted 2019-08-13 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity | interventions — Deoxycholic Acid

STUDY DESIGN:
Intervention Model Description: All subjects will receive deoxycholic acid (1-4 treatment sessions) for treatment of upper inner thigh fat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- deoxycholic acid (Experimental): Deoxycholic acid (Kybella) 10 mg/ mL will be injected subcutaneously, targeting the medial thigh deep fat compartment (pre-fascial). Subjects will receive deoxycholic acid 2 mg/ cm2, with injections of 0.2 mL spaced evenly 1 cm apart within the treatment area. Bilateral thighs will be treated. Each treatment will consist of a maximum of 8 mL (40 injection sites) of the study drug, with a maximum of 4 mL (20 injection sites) of the study drug for each thigh. Subjects will undergo 1-4 treatment sessions, each treatment session separated by 6 weeks +/- 1 week (Treatment #2, #3, or #4 will be pursued if patient desires more treatment, and if there is sufficient fat for treatment, per investigator's judgment.)
  Interventions: Drug: Deoxycholic Acid

INTERVENTIONS:
Drug: Deoxycholic Acid — Deoxycholic acid (Kybella) 10 mg/ mL subcutaneous

SUMMARY:
This is a phase I, open-label clinical trial evaluating the safety and efficacy of deoxycholic acid injection for reduction of upper inner thigh fat.

DETAILED DESCRIPTION:
Unwanted upper inner thigh fat is a common aesthetic complaint from patients, and current treatment options include liposuction and cryolipolysis (CoolSculpting, Allergan, Irvine, CA). Deoxycholic acid (Kybella, Allergan, Irvine, CA) is an FDA-approved injectable for the treatment of excess submental fat. At this time, it is not known if deoxycholic acid may be a safe and effective treatment for upper inner thigh fat. The proposed clinical trial will evaluate the safety and efficacy of deoxycholic acid for reduction of upper inner thigh fat.

In this single-arm, open-label safety and efficacy study, 15 subjects with excess upper inner thigh fat will receive 1-4 treatment sessions of subcutaneously injected deoxycholic acid. Subjects will be followed for 12 weeks after last treatment. Adverse events will be monitored. Efficacy will be objectively measured by change in thigh circumference; change in upper inner thigh skin fold thickness; increase in "thigh gap;" and percent accuracy by three blinded physicians in correctly identifying baseline photographs, upon independent review of before-and-after clinical photographs of the treatment area. Patient satisfaction related to the study treatment will be assessed with a Subject Self-Rating Scale throughout the study, and with a Post-Treatment Satisfaction Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 65
2. Discrete area of mild-to-moderate excess upper inner thigh fat, amenable to treatment at the discretion of the investigator
3. Subjects who score 0 (extremely dissatisfied) to 2 (slightly dissatisfied) on a Subject Self-Rating Scale, pertaining to upper inner thigh fat, with the scale ranging from 0 (extremely dissatisfied) to 6 (extremely satisfied)
4. Body mass index (BMI) less than 30 kg/m2
5. Stable body weight for previous 6 months (weight within 10 pounds of baseline)
6. Subjects must be in stable health, as confirmed by medical history, per investigator judgment
7. Subjects must be able to read, sign, and understand the informed consent
8. Subjects must we willing to avoid any other treatments to the inner thigh, including cryolipolysis and liposuction, during the study period.
9. Subjects must be willing to avoid changes in diet or exercise, any weight loss program, and any weight loss supplements, during the study period.
10. Subjects must be able and willing to avoid anticoagulation (aspirin, warfarin, heparin, rivaroxaban) for 1 week prior to each study treatment

Exclusion Criteria:

1. History of treatment for inner thigh fat, including cryolipolysis, noninvasive body contouring or liposuction in the last year
2. Previous trauma or surgery to pelvis or thighs
3. Subjects with an unstable medical condition, as deemed by the investigator
4. Women who are pregnant or lactating or plan to become pregnant during the study period
5. Lymphedema or edema of thigh
6. Excessive skin laxity in the treatment area, as judged by the investigator
7. Severe thigh cellulite
8. Subjects with any disease in the treatment area, such as dermatologic disease, that may be exacerbated by the study treatment
9. Subjects with any condition that may impair the evaluation of inner thigh fat
10. Subjects with known bleeding diathesis
11. Subjects with any known hypersensitivity to Kybella (deoxycholic acid) or any of the inactive ingredients: benzyl alcohol, dibasic sodium phosphate, sodium chloride, sodium hydroxide, hydrochloric acid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arisa Ortiz, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events pertaining to pre-assignment.
Period: Overall Study
Arm/Group | Deoxycholic Acid
Started | 15
Completed | 12
Not Completed | 3
Not completed — COVID | 3

BASELINE CHARACTERISTICS:
Arm/Group | Deoxycholic Acid
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 35 [22 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
BMI [Mean (Full Range); unit: kg/m^2] | 24 [19.7 to 29.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: 1. Any adverse event (AE) ascertained by patient report or physician evaluation
  2. One or more serious adverse events (SAE) as defined by CTCAEv4
  3. Adverse events leading to study drug discontinuation.
Time Frame: Baseline to 12 weeks after last treatment
Population: AE in number of participants
Measure: Number; unit: participants
Groups:
- Deoxycholic Acid: single arm study without comparison
Arm/Group | Deoxycholic Acid
Number analyzed (Participants) | 12
participants
  ransient subcutaneous nodules | 08
  injection-site urticaria | 01
  Temporary numbness | 02

2. Primary Outcome: Thigh Circumference Change
Description: change in thigh circumference as measured by tape measure
Time Frame: Baseline to 12 weeks after last treatment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Deoxycholic Acid
Number analyzed (Participants) | 12
cm
  average change from baseline at 4 week | -1.8 (0.5)
  average change from baseline at 12 week | -2.2 (0.6)

3. Primary Outcome: Upper Inner Thigh Skin Fold Thickness Change
Description: change in upper inner thigh skin fold thickness as measured by body fat calipers
Time Frame: Baseline to 12 weeks after last treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Deoxycholic Acid
Number analyzed (Participants) | 12
mm
  average change from baselineat 4 week | -7.3 (2.10)
  average change from baseline at 12 week | -8.8 (2.53)

4. Primary Outcome: Change in Thigh Gap
Description: Thigh gap," measured with a handheld soft ruler, was defined as the horizontal distance between baseline "sites of maximum bulge," with feet at standardized distance apart.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Deoxycholic Acid ?Placebo: Deoxycholic acid / Placebo
Arm/Group | Deoxycholic Acid ?Placebo
Number analyzed (Participants) | 12
centimeters | 1.6 (0.8)

5. Secondary Outcome: Percent Accuracy by Three Blinded Physicians in Correctly Identifying Before-and-after Photographs
Description: 3 blinded physicians identified the before and after photos and the percentage number was 83% for percent accuracy of the results. The percent accuracy was calculated for the entire Arm/Group rather than for each participant
Time Frame: 12 weeks
Measure: Number; unit: percent accuracy of post treatment photo
Arm/Group | Deoxycholic Acid
Number analyzed (Participants) | 12
percent accuracy of post treatment photo | 83

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire study duration (up to 12 weeks after last treatment, or up to 9 months).
Description: Does not differ from clinicaltrials.gov. since this is a local treatment with minimal to no systemic affects, there is no risk of mortality to subjects. Subjects may experience adverse events described in the study description.
Arm/Group | Deoxycholic Acid
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deoxycholic Acid (N=15)
pain (Skin and subcutaneous tissue disorders) | 15 (15)
swelling (Skin and subcutaneous tissue disorders) | 15 (15)
erythema (Skin and subcutaneous tissue disorders) | 15 (15)
bruising (Skin and subcutaneous tissue disorders) | 15 (15)

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, three subjects could not complete their 12-week follow-up visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT04054011/Prot_SAP_000.pdf